CLINICAL TRIAL: NCT05641480
Title: Technical R&D and Demonstration of Intelligent Medical Care in Alzheimer's Disease's Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaanxi Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020ZDLSF04-03
Record Dates: First submitted 2022-11-20; First posted 2022-12-07 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Alzheimer Disease; Subjective Cognitive Decline; Mild Cognitive Impairment; Mild Dementia
Keywords: Alzheimer's Disease; Subjective Cognitive Decline; Mild Cognitive Impairment; Mild Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Donepezil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjective cognitive decline group (Experimental): Studies suggest that acupuncture point Shenting can reduce the levels of serum inflammatory factors IL-6 and TNF-α, and the activity of cholinesterase of these two inflammatory factors is increased, and the activity of cholinacetylase is inhibited, which leads to brain tissue damage, nerve damage and cognitive dysfunction. Shenting（DU24）, Benshen（BG13） and Tou Wei（ST8） are the acupoints on the forehead, which have the effect of awakening the brain. Moreover, after acupuncture, nerve and periosteum effects can be caused, so as to improve cognitive function.
  Music therapy is a convenient and efficient method, and as a non-drug intervention, activate the memory to help people with Alzheimer's disease, trigger positive emotions, improve the symptoms of behavior, the moment of life in participants with Alzheimer's disease has great significance, is a good way to help participants with slow disease progression and improve the quality of life, increase happiness of life.
  Interventions: Device: Transcutaneous electrical acupoint stimulation&Music therapy
- Mild cognitive impairment group (Experimental): Studies suggest that acupuncture point Shenting can reduce the levels of serum inflammatory factors IL-6 and TNF-α, and the activity of cholinesterase of these two inflammatory factors is increased, and the activity of cholinacetylase is inhibited, which leads to brain tissue damage, nerve damage and cognitive dysfunction. Shenting（DU24）, Benshen（BG13） and Tou Wei（ST8） are the acupoints on the forehead, which have the effect of awakening the brain. Moreover, after acupuncture, nerve and periosteum effects can be caused, so as to improve cognitive function.
  Music therapy is a convenient and efficient method, and as a non-drug intervention, activate the memory to help people with Alzheimer's disease, trigger positive emotions, improve the symptoms of behavior, the moment of life in participants with Alzheimer's disease has great significance, is a good way to help participants with slow disease progression and improve the quality of life, increase happiness of life.
  Interventions: Device: Transcutaneous electrical acupoint stimulation&Music therapy
- Mild dementia group (Experimental): On the basis of the above two treatment options, oral donepezil hydrochloride tablets or carpalatine heavy tartrate tablets should be added.
  Interventions: Drug: Donepezil hydrochloride tablets or carpalatine bitartrate tablets

INTERVENTIONS:
Device: Transcutaneous electrical acupoint stimulation&Music therapy — Procedure: electro-acupuncture;Points: Shenting（DU24）, Benshen（BG13）, Tou Wei （ST8）.The specially-made pad is stick on pierced acupoints, until local sour and heavy feeling coming. The electric stimulator is applied to bilateral BG13 and ST8, with dilatational wave,10/50 Hz and electric current 1-5mA(milliampere).Every session lasts for 30 min per day. The participants are treated continuously for 8 weeks for 3 sessions a week, 24 sessions for each participants in all.
  Selecting the participants' music of memory and music of favourite(Music is purchased and downloaded from music stores), forming a personalized music playlist, and the decibel level is suitable for participants.
  The treatment is designed based on recent literature research in 10 years, former result and expert consensus.
  Other Names:
  * JS-502-A Intelligent and portable electroacupuncture
  * apparatus(Han's low frequency neuromodulator, made in China)
  Arms: Mild cognitive impairment group; Subjective cognitive decline group
Drug: Donepezil hydrochloride tablets or carpalatine bitartrate tablets — ① Donepezil hydrochloride tablets 5 mg, once a day, one tablet each time, before going to bed. The treatment period is 6 months.
  ② Carpalatine heavy tartrate tablets 1.5mg, 1 tablet/time 2 weeks before treatment, twice a day, breakfast and dinner with food, swallow. If there is no obvious adverse reaction after 2 weeks, the dosage can be increased to 2 tablets/time, twice a day. The treatment period is 6 months.
  Arms: Mild dementia group

SUMMARY:
This is a study on patient registry, and the sample size of this clinicaltrial is designed in group sequential design. According to the diagnostic criteria, the subjects are divided into SCD group, MCI group and mild dementia group. At the early stage of treatment, the investigators give participants transcutaneous electrical acupoint stimulation and music therapy according to the guidance of TCM syndrome differentiation. Participants can treat themselves at home after the investigators give them intelligent device and music，and according to the TCM syndrome score, neuropsychological scale, curative effect evaluation of daily life ability scale, determining the optimal comprehensive treatment plan,and phase in the treatment of participants with food, clothing, shelter, line, and life aspects of health education and guidance, a total of 24 weeks of treatment.

DETAILED DESCRIPTION:
As China progresses toward an aging society, the prevalence of geriatric diseases increases with it, especially in the case of Alzheimer's Disease (AD), the main clinical features of which are memory loss, cognitive dysfunction and behavioral impairment. At present, the disease is the fourth cause of death in the world after heart disease, tumor and stroke, which seriously causes heavy economic and social burden. Because the etiology of AD is not clear and the pathogenesis is complex, there is still a lack of effective treatment to curb its progress.

This project focuses on alzheimer's disease, according to the law of development for a disease to occur, combined with traditional Chinese medicine theory, the investigators according to the guidance of syndrome differentiation for participants with percutaneous acupoint stimulation and music therapy intervention plan.Mild dementia participants increase donepezil hydrochloride tablets or carbalatine bitartrate tablets. The therapeutic effect is evaluated once at 4 weeks and 8 weeks during the treatment period, and once at 12 weeks and 24 weeks during the follow-up period, a total of 4 times. After the treatment, the number of cases with stable condition, the number of cases with normal condition and the number of cases with disease transformation are calculated according to the diagnostic criteria. The efficacy and caregiver burden are evaluated according to dementia syndrome scale and neuropsychological scale.

In recent years, traditional Chinese medicine (TCM) has been expanding in the field of AD research. The individualized treatment methods of syndrome differentiation and treatment, as well as the multi-target and multi-means intervention techniques have obvious curative effects on improving cognitive status and delaying the progression of the disease, without obvious side effects and adverse reactions.Acupoint stimulation methods, such as acupuncture, warm moxibustion, acupoint application, electrical stimulation are all used to dredge human meridians to adjust the spirit, strengthen the brain and improve cognitive function. Therefore, the above comprehensive TCM intervention program may be the key link in the early prevention and treatment of AD.

This is a study on patient registry, and the sample size of this clinicaltrial is designed in group sequential design. According to the diagnostic criteria, the subjects are divided into SCD group, MCI group and mild dementia group. At the early stage of treatment, the the investigators give participants transcutaneous electrical acupoint stimulation and music therapy according to the guidance of TCM syndrome differentiation. Participants can treat themselves at home after the investigators give them intelligent device and music，and according to the TCM syndrome score, neuropsychological scale, curative effect evaluation of daily life ability scale, determining the optimal comprehensive treatment plan,and phase in the treatment of participants with food, clothing, shelter, line, and life aspects of health education and guidance, a total of 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria of SCD, MCI and mild dementia;
* Memory decline (self-reported or confirmed by both informants);
* Age 55-75 years;
* Memory impairment has not reached the diagnostic criteria of moderate and severe dementia;
* Hachinski ischemia scale score ≤ 4;
* Exclude any other systemic diseases that can cause brain dysfunction;
* Hamilton Depression Scale < 17;
* The subject or guardian signed the informed consent.

Exclusion Criteria:

* There are advanced, serious or unstable other diseases, such as liver, kidney and other serious primary diseases;
* Severe hearing and visual impairment, can not cooperate with the assessment;
* with active epilepsy;
* Previous history of mental illness;
* Moderate or severe dementia, cerebral infarction or any physical or mental disorder that may lead to brain dysfunction;
* Having used other drugs that may cause cognitive function changes or heart, brain, kidney and other important organs failure before inclusion;
* Under 55 years old or above 75 years old;
* Unable to cooperate with the completion of the corresponding assessment and inspection and quit;
* Those who are likely to have poor compliance with the test;
* Participants in other subjects.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2025-12-09 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
AD-seeds protein analyzer（Developed by Professor Jia Jianping of Capital Medical University of China） | Change from Baseline Aβ level at 6 months
  The area under curve is used to show the ability of the AD-seeds-detector to diagnose AD. The value of area under curve is higher, then the ability of the AD-seeds-detector to diagnose AD is stronger.AD-seeds protein analyzer is an antibody-free and cost-efective approach for measuring blood biomarkers. It's a newly developed instrument to distinguish Alzheimer's disease (AD) from other forms of dementia.It examines amyloid in the blood. Alzheimer's disease is usually not discovered until the late stage, and early detection and intervention are of great significance to improve the treatment effect of the disease.
Or adopting Serum Aβ level is detected | Change from Baseline Aβ level at 6 months
  A certain amount of fasting venous blood is collected from participants before and after treatment, and the supernatant is collected by low-speed centrifugation at a certain temperature. The serum Aβ level is detected by enzyme-linked immunosorbent assay (ELISA)

SECONDARY OUTCOMES:
Electrocardiogram（ECG） | Change from Baseline at 6 months（Week -1~0 day, week 24 ± 3 days）
  ECG QT Interval.（Security Index）
Change of total MMSE score from baseline | Change from Baseline at 6 months（FIve times：Week -1~0 day，Week 4 ± 2 days，week 8 ± 2 days，week 12 ± 3 days，week 24 ± 3 days）
  MMSE score are commonly used for estimating the severity of cognitive impairment with maximum score of 30. The questions in this scale included orientation to time, orientation to place, attention and calculation, recall of three words and visual construction.It can comprehensively, accurately and rapidly reflect the degree of mental state and cognitive impairment of the subjects. To provide scientific basis for clinical psychological diagnosis, treatment and neuropsychological research.
Montreal Cognitive Assessment Scale (MoCA) Score | Change from Baseline at 6 months（FIve times：Week -1~0 day，Week 4 ± 2 days，week 8 ± 2 days，week 12 ± 3 days，week 24 ± 3 days）
  MoCA is an assessment tool used for rapid screening of abnormal cognitive function, including 11 examination items in 8 cognitive fields, with a total score of 30 points, among which a score ≥26 is considered as normal cognitive function. Its high sensitivity, covering important cognitive fields, short test time, suitable for clinical application. The MoCA scores of the two groups are recorded before and after treatment.
Disease conversion rate A | Baseline，6 months
  The disease conversion rate is calculated to evaluate the application effect of this model in elderly people with cognitive dysfunction.The number of stable dementia cases is calculated according to the diagnostic criteria of dementia symptom staging.
Disease conversion rate B | Baseline，6 months
  According to the diagnostic criteria of dementia symptom staging, the number of participants turned to normal is calculated.
Disease conversion rate C | Baseline，6 months
  According to the diagnostic criteria of dementia symptom staging, the number of disease conversion cases is calculated.
Disease conversion rate D | Baseline，6 months
  The conversion of SCD to MCI/ Alzheimer's disease is calculated according to the diagnostic criteria of dementia symptom staging.
Disease conversion rate E | Baseline，6 months
  According to the diagnostic criteria of dementia symptom staging, MCI is converted to Alzheimer's disease.
Disease conversion rate F | Baseline，6 months
  According to the diagnostic criteria of dementia symptom staging, the conversion rate of mild dementia to moderate to severe dementia is calculated.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shaanxi Hospital of Traditional Chinese Medicine,, Xi'an, Shaanxi
  - Shaanxi Hospital of Traditional Chinese Medicine, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR